CLINICAL TRIAL: NCT07329296
Title: The Regenerative Capacity of the Donor Liver After Living Donor Liver Transplantation: an Ambidirectional Cohort Study
Acronym: LRLDLT
Status: Enrolling by invitation | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Robert Minnee, MD, PhD, Erasmus Medical Center
Other Study IDs: MEC-2025-0362
Record Dates: First submitted 2025-12-29; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Living Donor Liver Transplantation
Keywords: Liver Transplantation; Living Donor; Magnetic Resonance Imaging; Liver Regeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Living liver donors: The population consists of adult living liver donors at the Erasmus MC.
  Interventions: Procedure: Living liver donation

INTERVENTIONS:
Procedure: Living liver donation — Adults who underwent living liver donation.

SUMMARY:
Rationale: Living donor liver transplantation (LDLT) offers a promising solution to the organ shortage. During living liver donation, a substantial portion of the donor's liver is resected. Fortunately, the liver has a remarkable capacity to regenerate. However, liver regeneration varies among individuals. Previous studies have identified several clinical factors as potential predictors of regenerative capacity. Nevertheless, these studies are outdated and do not reflect current clinical practice or recent advancements. This study aims to investigate the regenerative capacity of the donor liver following LDLT and identify its clinical predictors. It is hypothesized that the liver regenerates to the original size.

Objectives: The main objective of this study is to evaluate the regenerative capacity of the donor liver following LDLT. The secondary objective is to identify clinical predictors of the regenerative capacity of the donor liver following LDLT.

Study type: This is an ambidirectional, single-center cohort study using medical records.

Study population: The population consists of adult living liver donors aged 18-60 years at the Erasmus MC who donate(d) between May 2004 and June 2026 and gave written informed consent.

Methods: General, graft weight and liver volumetry data will be extracted from HiX. The study coordinator will register his findings and analyze them. The paired samples t-test will be used to test for differences in mean remnant liver volume and liver volume 12 months post-donation. In addition, subgroup analyses will be performed for sex, age, weight, type of liver graft donation, anatomical variants, liver steatosis, and donor complications. Multiple linear regression analysis will be performed for sex, age, BMI, donor length of stay, remnant liver volume and percentage, and type of liver graft donation.

DETAILED DESCRIPTION:
Research methods: General and graft weight data will be extracted from HiX. Additionally, liver volume pre-donation (VPRD) and 12 months post-donation (V12M) from CT- or MRI-volumetry will be extracted from HiX. The study coordinator will register his findings in Castor.

Analysis: Normality will be tested using the Shapiro-Wilk test. Homogeneity of variances will be tested using the F-test. A QQ plot will be used to check for outliers. For the baseline donor characteristics, mean (standard deviation (SD)) age, weight, height, BMI, and the percentage of females and related donations, will be calculated. A table of these parameters will be made.

The surgical outcomes OR time, blood loss, donor LOS, and Clavien-Dindo ≥III complications will be described and mean (SD) of these parameters will be calculated. A table of these parameters will be made.

The mean (SD) remnant liver volume (RLV) and V12M will be calculated. The regenerative capacity will be calculated by the formula: regenerative capacity = V12M/RLV * 100(%). For the mean regenerative capacity, the average of all donors' regenerative capacities will be taken. A table showing the means (SD) and min-max of RLV, V12M, and the regenerative capacities will be made. The distribution of regenerative capacities will be shown in a bar chart. The paired samples t-test will be used to test for differences in mean RLV and liver volume 12 months post-donation (V12M). In addition, subgroup analyses will be performed for sex, age (<40 vs ≥40 years), weight (<70 vs ≥70 kg), type of liver graft donation (right vs left lobe), anatomical variants, liver steatosis, and donor complications using the unpaired samples t-test, Welch's t-test, or Mann-Whitney test. Multiple linear regression analysis will be performed for the following 7 potential predictors of regenerative capacity: sex, age, BMI, donor LOS, remnant liver volume and percentage, and type of liver graft donation (right vs left lobe). Variance inflation factor (VIF) will be used to test for multicollinearity. Statistical analyses will be carried out using RStudio 2024.09.1, GraphPad Prism 9.5.0, and Microsoft Excel version 16.90.2. P<0.05 indicates statistical significance.

Recruitment and informed consent procedures: The transplant coordinator and/or transplant surgeon will inform participants about the study and will ask their written informed consent. Living liver donors are followed up annually for life. The participants will be informed during a follow-up consult. All donors who are, for whatever reason, not visiting the Erasmus MC anymore for follow-up are contacted by phone. If the donor considers participating, a Patient Information Form (PIF) will be sent by mail. The donors can return the signed PIF through mail. Donors can withdraw their informed consent at any time and for any reason if they wish to do so without any consequences. They can withdraw through phone, mail, or in person.

Privacy protection: Subject's privacy is protected by using coded data. In the database subjects are referred to as numbers. These numbers are chosen at random. Which number belongs to which subject is registered in a key table with a password. This password is only known by the principal investigator and the research team. The database in which the data is stored (Castor), meets the requirements set for data security. The handling of personal data is in compliance with the Dutch Data Protection Act (in Dutch: 'Algemene Verordening Gegevensbescherming (AVG)). Only the code number will be used for study documentation, progress reports, and research publications.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* Living liver donation between May 2004 and June 2026
* Written informed consent

In order to be eligible for LDLT, a subject needed to meet all of the following criteria:

* 18-60 years old
* Physical and mental well-being
* Body Mass Index (BMI) <33 kg/m2
* No active drugs or other substances use

Exclusion Criteria:

There are no exclusion criteria for this study.

Exclusion criteria for LDLT were:

Absolute exclusion criteria

* Medical conditions (for instance heart disease and bleeding or clotting disorders)
* History of liver disease
* Previous/active malaria infection
* Financial incentive or indications of pressure
* Unable to cooperate with designated long-term follow-up
* Severe psychiatric disease or psychological instability
* Active alcoholism or frequent heavy alcohol use or drugs use/abuse
* Unable to give informed consent
* History of dementia or other neurological degenerative disorders
* Persons with rabies or persons bitten in the past 6 months by an animal and that are treated as if the animal is rabid
* Persons with syphilis
* Human immunodeficiency virus-positive persons. Relative exclusion criteria
* BMI >33 kg/m2
* Smoking

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The population consists of adult living liver donors at the Erasmus MC.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Liver regeneration | Preoperative during screening for living liver donation and 1 year post-donation.
  The primary outcomes are remnant liver volume (RLV), assessed by subtracting the graft weight from the volume pre-donation, and the liver volume 12 months post-donation. Liver volumes are assessed with CT- or MRI-volumetry.

SECONDARY OUTCOMES:
Predictors | Preoperative during screening for living liver donation and during follow-up until 1 year post-donation.
  Secondary outcomes are clinical parameters possibly correlated with the regenerative capacity of the donor liver after LDLT. The following clinical predictors are studied: gender, age, BMI, donor length of stay, remnant liver volume and percentage, type of liver graft donation (right vs left lobe), anatomical variants, and liver steatosis.

CONTACTS AND LOCATIONS:
Overall Officials: Robert C. Minnee, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, documentation, data management plan, data analysis plan, script to assess data, scripts to analyse data, scripts to generate tables and figures in the publication.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: (Underlying) data will be made available alongside with the publication. It will be available for 10 years. Access to the data and images is approved by the head of department and principal investigator. This access is temporarily. To whom and when access approved is registered.
Access Criteria: The PI will verify the authenticity of the requesting researcher and will check whether their intentions are in line with the informed consent and whether the intended methodology is suitable and will approve the request before providing access to the data. Other researchers could express their interest in the dataset through countersigned DTA. After meeting the sharing and reuse conditions as described above and approval of the PI, data access will be provided through the data repository.

REFERENCES:
- [Background] Pomfret EA, Pomposelli JJ, Gordon FD, Erbay N, Lyn Price L, Lewis WD, Jenkins RL. Liver regeneration and surgical outcome in donors of right-lobe liver grafts. Transplantation. 2003 Jul 15;76(1):5-10. doi: 10.1097/01.TP.0000079064.08263.8E. PMID 12865779
- [Background] Michalopoulos GK. Liver regeneration. J Cell Physiol. 2007 Nov;213(2):286-300. doi: 10.1002/jcp.21172. PMID 17559071
- [Background] Yim SH, Kim DG, Kang M, Koh HH, Choi MC, Min EK, Lee JG, Kim MS, Joo DJ. Survival benefit of living-donor liver transplantation in patients with a model for end-stage liver disease over 30 in a region with severe organ shortage: a retrospective cohort study. Int J Surg. 2023 Nov 1;109(11):3459-3466. doi: 10.1097/JS9.0000000000000634. PMID 37565633